CLINICAL TRIAL: NCT01488240
Title: The Role of Pulsed Dye Laser Therapy in the Management of Burn Scars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B2011: 074
Record Dates: First submitted 2011-12-05; First posted 2011-12-08 (Estimated); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Burn Scar
Keywords: burn; scar; laser
MeSH Terms: conditions — Burns; Cicatrix | interventions — Lasers, Dye

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Proximal (Active Comparator): part of scar proximal to heart
  Interventions: Procedure: pulsed dye laser
- Distal (Active Comparator): part of scar distal to heart
  Interventions: Procedure: pulsed dye laser

INTERVENTIONS:
Procedure: pulsed dye laser — laser energy

SUMMARY:
The purpose of this study is to determine the effects (good or bad) of pulsed dye laser treatment in burn scar height, texture, redness and pliability in acute burn injury.

DETAILED DESCRIPTION:
While the literature tends to support the use of laser therapy in the management of burn scars, there is a definite lack of appropriately powered, randomized controlled trials. Laser therapy can be quite expensive when compared to other treatment modalities for burn scars, and while promising, its true usefulness has yet to be conclusively demonstrated. For this reason, our research group is proposing the commencement of two randomized controlled trial pilot studies assessing the effects of pulsed dye laser (PDL) on burn scars. The objectives of this project will be to determine the effectiveness of pulsed dye laser therapy on burn scar vascularity, pliability, height and texture. It has been hypothesized that the PDL works on acute injury to decrease scar formation, and the fractional laser works on scar that is quiescent to promote remodelling. Therefore the investigators are proposing to study both acute injury and late burn scars. This project will compare the effects of each laser type, and will either help support or refute the assertion that laser therapy can be used to improve burn scars.

Objectives:

To determine the benefit of pulsed dye laser treatment in improving burn scar height, texture, vascularity and pliability in acute burn injury.

ELIGIBILITY:
Inclusion Criteria:

* burn scar
* living in Winnipeg
* scar age one to 6 months
* Fitzpatrick I-III skin type

Exclusion Criteria:

* open wound
* active infection
* previous scar treatment with steroid injection or interferon
* established disposition towards keloid scarring

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2012-11-01; Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Scar Characteristics | six months
  Examine characteristics of scar

CONTACTS AND LOCATIONS:
Overall Officials: S Logsetty, MD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada